CLINICAL TRIAL: NCT01307904
Title: The Glycemic Indices of Five Common Varieties of Dates in the Tested Among Healthy and Diabetic Subjects
Acronym: Dates
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Collaborators: Abu Dhabi Food Control Authority (Other Government)
Responsible Party: Juma M Alkaabi, Faculty of Medicine and Health Sciences - UAE University
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: UAEU Dates GI Study
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus
Keywords: Glycemic index; Dates; Blood glucose
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose; Chronology as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dates (Active Comparator): Each healthy and diabetic subjects received 50 grams equivalent of carbohydrates of the tested dates, On five separate days.
  Interventions: Other: Dates
- sugar (Active Comparator): Each healthy and diabetic subjects received 50 grams of glucose
  Interventions: Other: Glucose

INTERVENTIONS:
Other: Glucose — Each healthy and Diabetic volunteers received 50 grams of glucose
  Arms: sugar
Other: Dates — Each healthy and diabetic volunteers received 50 grams equivalent of carbohydrates of each of the five selected dates, on five separate days.
  Arms: dates

SUMMARY:
The main objectives of this study is to measure the composition of five common types of dates (Fara'd, Lulu, Abu ouma'n, Dabbas and Khalas) and to calculate their Glycemic Indices (GI) of these dates tested in healthy and diabetic subjects. Thirteen healthy volunteers and ten subjects with type 2 diabetes mellitus were enrolled in the study.

The dates' flesh composition analysis showed that the dates contain a high percentage of carbohydrate (total sugars, 65-68%).

The measured mean glycemic indices of the dates among healthy individuals were 54.0, 53.5, 46.3, 49.1 and 55.1 for Fara'd, Lulu, Abu Ouma'n, Dabbas and Khalas, respectively. Corresponding mean glycemic indices among individuals with type 2 diabetes were very similar 46.1, 43.8, 51.8, 50.2, and 53.0. Thus the tested five varieties of the dates are classified as low glycemic index food items.

DETAILED DESCRIPTION:
The United Arab Emirates (UAE) has transitioned rapidly over the last 40 years. This has lead to a dramatic increase in the prevalence of obesity, metabolic syndrome, dyslipidaemia, hypertension, prediabetes and diabetes. Daily consumption of dates is the norm.The main objectives of this study is to measure the composition of five common types of dates (Fara'd, Lulu, Abu ouma'n, Dabbas and Khalas) and to calculate their Glycemic Indices (GI) of these dates tested equally in healthy and diabetic subjects. Thirteen healthy volunteers and ten subjects with type 2 diabetes mellitus were enrolled in the study. The dates' flesh composition analysis showed that the dates contain a high percentage of carbohydrate (total sugars, 65-68%).

The measured mean glycemic indices of the dates among healthy individuals were 54.0, 53.5, 46.3, 49.1 and 55.1 for Fara'd, Lulu, Abu Ouma'n, Dabbas and Khalas, respectively. Corresponding mean glycemic indices among individuals with type 2 diabetes were very similar 46.1, 43.8, 51.8, 50.2, and 53.0. Thus the tested five varieties of the dates are classified as low glycemic index food items with potential health benefits for healthy and diabetic individuals alike.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Healthy or having controlled type 2 diabetes mellitus

Exclusion Criteria:

* Morbid obesity (BMI > 40)
* Presence of gastroenterological disorders
* Alimentary tract surgery
* A history of gastroenteritis in the prior six months
* Any disease that may affect glucose metabolism
* Alcohol intake
* Smoking
* Taking any medications (except metformin)
* Poorly uncontrolled diabetes (HbA1c > 8%)
* The presence of chronic diseases or the presence of acute illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Dates Glycemic Index | 4 months
  Measuring the composition of dates, selection of patients and carrying out the study

CONTACTS AND LOCATIONS:
Overall Officials: Juma M Alkaabi, MD, Principal Investigator — Faculty of Medicine and Health Sciences, UAE University; Bayan Al-Dabbagh, PhD, Study Director — Faculty of Medicine and Health Sciences, UAE University; Professor Hussein saadi, MD, Study Director — Faculty of Medicine and Health Sciences, UAE University; Professor Salah Gariballa, FRCP, Study Director — Faculty of Medicine and Health Sciences, UAE University; Ahmed Shakeel, PhD, Study Director — Abu Dhabi Food Control Authority; Mustafa Al Gazali, PhD, Study Director — Abu Dhabi Food Control Authority
Locations (1):
- Internal Medicine Department, FMHS, UAE University, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

REFERENCES:
- [Derived] Alkaabi JM, Al-Dabbagh B, Ahmad S, Saadi HF, Gariballa S, Ghazali MA. Glycemic indices of five varieties of dates in healthy and diabetic subjects. Nutr J. 2011 May 28;10:59. doi: 10.1186/1475-2891-10-59. PMID 21619670